CLINICAL TRIAL: NCT01362972
Title: Analysis of Data Collected in the European Group for Blood and Marrow Transplantation (EBMT) Registry on a Cohort of Patients Receiving Plerixafor
Status: Completed | Type: Observational
Sponsor: Genzyme, a Sanofi Company (Industry)
Collaborators: European Society for Blood and Marrow Transplantation (Network)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: MOZ18009; OBS13611 (Other: Sanofi)
Record Dates: First submitted 2011-05-27; First posted 2011-06-01 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Lymphoma; Multiple Myeloma
MeSH Terms: conditions — Lymphoma; Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- plerixafor + granulocyte colony stimulating factor (G-CSF): Patients who receive plerixafor+granulocyte colony stimulating factor (G-CSF) for the mobilisation of peripheral blood (PB) CD34+ cells and who have undergone autologous haematopoietic stem cell (HSC) transplantation.
- plerixafor + G-CSF + chemotherapy: Patients who receive plerixafor+granulocyte colony stimulating factor (G-CSF)+chemotherapy for the mobilisation of peripheral blood (PB) CD34+ cells and who have undergone autologous haematopoietic stem cell (HSC) transplantation.
- granulocyte colony stimulating factor (G-CSF) + chemotherapy: Patients who receive granulocyte colony stimulating factor (G-CSF) + chemotherapy for the mobilisation of peripheral blood (PB) CD34+ cells and who have undergone autologous haematopoietic stem cell (HSC) transplantation.
- granulocyte colony stimulating factor (G-CSF) alone: Patients who receive granulocyte colony stimulating factor (G-CSF) alone for the mobilisation of peripheral blood (PB) CD34+ cells and who have undergone autologous haematopoietic stem cell (HSC) transplantation.

SUMMARY:
In the European Union (EU), plerixafor is indicated in combination with granulocyte colony stimulating factor (G-CSF) to enhance mobilisation of haematopoietic stem cells (HSCs) to the peripheral blood (PB) for collection and subsequent autologous transplantation in patients with lymphoma and multiple myeloma (MM) whose cells mobilise poorly.

This is a clinical outcome analysis of a prospectively defined cohort of patients with data reported retrospectively to the European Group for Blood and Marrow Transplantation (EBMT) who have lymphoma or multiple myeloma (MM), whose cells mobilize poorly, and who have undergone autologous haematopoietic stem cell (HSC) transplantation during the years 2008 up to and including 2012.

The EBMT is a non-profit, scientific society representing more than 600 transplant centers mainly in Europe. The EBMT promotes all activity aiming to improve stem cell transplantation or cellular therapy, which includes registering all the activity relating to stem cell transplants. Data are entered, managed, and maintained in a central database with internet access; each EBMT center is represented in this database.

The analysis of data from a well established registry like the EBMT registry allows for follow up of a large number of patients who are representative of the patient population receiving plerixafor.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the cohort analysis, patients must have data in the EBMT registry that meet the following criteria:

* Adults diagnosed with lymphoma or multiple myeloma (MM)
* Received first autologous transplants of peripheral blood (PB) non ex-vivo manipulated stem cells in the time period listed above using cells mobilised with one of the following regimens:

  * plerixafor plus granulocyte colony stimulating factor (G-CSF)
  * plerixafor plus G-CSF plus chemotherapy
  * G-CSF alone or
  * G-CSF plus chemotherapy

Note: Patients included in the plerixafor groups will be those treated according to the label

* Provision of informed consent (i.e., all patients with data in the EBMT registry will have signed consent at the time of transplantation for the potential use of their data for analysis)

Exclusion Criteria:

* Patients treated with plerixafor NOT according to the European Union (EU) label.
* Patients whose graft product underwent ex vivo manipulation will be excluded from analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with data reported to the EBMT who have lymphoma or multiple myeloma (MM) and who have undergone autologous haematopoietic stem cell (HSC) transplantation during the years 2008 up to and including 2012.
Sampling Method: Non-Probability Sample
Enrollment: 7801 (Actual)
Dates: Start 2011-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Compare PFS, OS, and Relapse in EBMT-registered autoHSC transplant patients between 2008 and 2012, with HSCs mobilized with Plerixafor + G-CSF vs other regimens. | 5 Years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company

REFERENCES:
- [Derived] Sureda A, Chabannon C, Masszi T, Pohlreich D, Scheid C, Thieblemont C, Wahlin BE, Sakellari I, Russell N, Janikova A, Dabrowska-Iwanicka A, Touzeau C, Esquirol A, Jantunen E, van der Werf S, Bosman P, Boumendil A, Liu Q, Celanovic M, Montoto S, Dreger P. Analysis of data collected in the European Society for Blood and Marrow Transplantation (EBMT) Registry on a cohort of lymphoma patients receiving plerixafor. Bone Marrow Transplant. 2020 Mar;55(3):613-622. doi: 10.1038/s41409-019-0693-z. Epub 2019 Sep 30. PMID 31570781
- [Derived] Morris C, Chabannon C, Masszi T, Russell N, Nahi H, Kobbe G, Krejci M, Auner HW, Pohlreich D, Hayden P, Basak GW, Lenhoff S, Schaap N, van Biezen A, Knol C, Iacobelli S, Liu Q, Celanovic M, Garderet L, Kroger N. Results from a multicenter, noninterventional registry study for multiple myeloma patients who received stem cell mobilization regimens with and without plerixafor. Bone Marrow Transplant. 2020 Feb;55(2):356-366. doi: 10.1038/s41409-019-0676-0. Epub 2019 Sep 18. PMID 31534192
- [Derived] Auner HW, Iacobelli S, Sbianchi G, Knol-Bout C, Blaise D, Russell NH, Apperley JF, Pohlreich D, Browne PV, Kobbe G, Isaksson C, Lenhoff S, Scheid C, Touzeau C, Jantunen E, Anagnostopoulos A, Yakoub-Agha I, Tanase A, Schaap N, Wiktor-Jedrzejczak W, Krejci M, Schonland SO, Morris C, Garderet L, Kroger N. Melphalan 140 mg/m2 or 200 mg/m2 for autologous transplantation in myeloma: results from the Collaboration to Collect Autologous Transplant Outcomes in Lymphoma and Myeloma (CALM) study. A report by the EBMT Chronic Malignancies Working Party. Haematologica. 2018 Mar;103(3):514-521. doi: 10.3324/haematol.2017.181339. Epub 2017 Dec 7. PMID 29217776